CLINICAL TRIAL: NCT04384094
Title: Rebound Esthesiometer Phase 2 Protocol
Brief Title: Defining the Operating Parameters for a Rebound-esthesiometer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Icare Finland Oy (Industry)
Responsible Party: Sponsor
Other Study IDs: TE0X_EST_2
Record Dates: First submitted 2020-05-04; First posted 2020-05-12 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-04

CONDITIONS: Corneal Sensation Reduced; Corneal Dystrophy; Corneal Degeneration; Corneal Transplant Failure; Herpetic Keratitis
Keywords: esthesiometry; corneal sensitivity
MeSH Terms: conditions — Corneal Dystrophies, Hereditary; Keratitis, Herpetic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test subjects: Test subjects according to the inclusion / exclusion criterias.
  Interventions: Device: Esthesiometer measurement

INTERVENTIONS:
Device: Esthesiometer measurement — Measuring the corneal sensitivity using rebound technology.

SUMMARY:
The purpose of this study is to define the operating parameters for a new method to measure corneal sensitivity.

DETAILED DESCRIPTION:
Corneal sensitivity is the most important protective mechanism of the eye. Thus, measuring it at any given time gives important indicators of corneal physiology, especially in the diagnostics of corneal and systemic diseases (e.g. diabetes, herpes simplex and keratitis) and recovery from ocular surgery. Current commercial measurement methods are outdated, non-quantitative and uncomfortable to use, hence left unused. This results in suboptimal, even poor, diagnosis and treatment for patients.

In this study the operating parameters for a state-of-the-art esthesiometer are defined. The operating principle is based on existing rebound technology which is already approved for IOP measurement.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Informed consent signed

Exclusion Criteria:

* Signs of infectious or inflammatory disease of anterior eye at the time of presentation.
* During last two weeks, any of the following events or conditions occurred or was present: inflammatory or infectious ocular condition, surgical or other intervention or therapy, other abnormal ocular event.
* Unable to give informed consent.
* Directly or indirectly indicated vunerability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects entering ocular primary care examination site and patients entering eye hospital for several medical reasons.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Rebound esthesiometer operating threshold | 2020-2021
  Define the corneal touch sensitivity threshold using the rebound esthesiometer by varying the measurement probe impact at the moment of touch of corneal surface. The impact is varied by changing the speed (m/s) of the measurement probe and the subjective sensation of the test subject is recorded. The mass (mg) of the measurement probe is known and the impact energy is calculated.
Rebound esthesiometer operating parameters | 2020-2021
  Measure the correlation of corneal touch sensitivity between rebound esthesiometer and the reference instrument Cochet-Bonnet monofilament esthesiometer. With the rebound esthesiometer the impact is varied by changing the speed (m/s) of the measurement probe. The probe mass (mg) and speed (m/s) equals to the touch impact impulse which causes the touch sensation. The subjective sensation of the test subject is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Matjaz Mihelcic, Ph.D., Principal Investigator — Optika Mesec

IPD SHARING:
Plan to Share IPD: No